CLINICAL TRIAL: NCT00053196
Title: Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation For Patients With Disease Relapse Or Myelodysplasia After Prior Autologous Transplantation
Brief Title: Donor Stem Cell Transplant in Treating Patients With Relapsed Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-100002; U10CA031946 (NIH); CALGB-100002; CDR0000269301 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myeloproliferative Neoplasms
Keywords: refractory chronic lymphocytic leukemia; prolymphocytic leukemia; recurrent adult Hodgkin lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; previously treated myelodysplastic syndromes; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; atypical chronic myeloid leukemia, BCR-ABL negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Leukemia, Myeloid, Acute; Dendritic Cell Sarcoma, Interdigitating; Recurrence; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Antilymphocyte Serum; Granulocyte Colony-Stimulating Factor; Filgrastim; Busulfan; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Tacrolimus; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non myeloblative allogeneic transplant (Experimental): Non myeloblative allogeneic hematopoietic cell transplantation after prior autologous transplantation
  Interventions: Biological: anti-thymocyte globulin; Biological: G-CSF; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: allogeneic cell transplantation; Drug: allopurinol

INTERVENTIONS:
Biological: anti-thymocyte globulin — 2.5mg/kg/day IV infusion over 6 hrs x 4 doses Days -4 to -1 (for MUD and 9/10 related donor transplants only)
Biological: G-CSF — 5 ug/kg/day subQ injection Day 7 until ANC> 1000/uL for 3 consec days
  Other Names: filgrastim
Drug: busulfan — 0.8mg/kg IV infusion over 2 hrs q 6 hrs x 8 doses Days -4 thru -3
Drug: fludarabine phosphate — 30 mg/sq m/day IVBP over 30 min Days -7 thru -3
Drug: methotrexate — 5 mg/sq m/day IV infusion Days 1, 3, & 6 for HLA-identical donor transplants and Days 1, 3, 6, & 11 for MUD & 9/10 related donor transplants
Drug: mycophenolate mofetil — 15mg/kg PO bid Day -2 to Day 60, then taper as tolerated (for MUD and 9/10 related donor transplants only)
Drug: tacrolimus — target serum level is 5-10 ng/mL. Start with 0.03mg/kg PO bid Day -1 to Day 90, then taper thru Day 150 for HLA identical donor transplants and Day -1 to Day 180 then taper for MUD and 9/10 related donor transplants
Procedure: allogeneic cell transplantation — 2,000,000-8,000,000 CD34+ cells total via infusion Days 0 and 1
Drug: allopurinol — 300 mg/day PO Days -8 thru -1

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and busulfan, before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving immunosuppressive therapy after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor bone marrow or peripheral stem cell transplant works in treating patients with relapsed hematologic cancer after treatment with chemotherapy and autologous stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of non-myeloablative allogeneic hematopoietic stem cell transplantation by demonstrating that the risk of treatment-related mortality during the first 6 months is an acceptable rate of less than 40% in patients with relapsed hematologic malignancies after prior high-dose chemotherapy and autologous stem cell transplantation.
* Determine the response rates (disease-specific partial and complete response) in patients treated with this regimen.
* Determine the 6-month and 12-month probabilities of response in patients treated with this regimen.
* Determine the distribution of time-to-progression in patients responding to this regimen.
* Determine the percent donor chimerism in patients treated with this regimen.
* Determine the risk of acute and chronic graft-vs-host disease in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the disease-free and overall survival of patients treated with this regimen.

OUTLINE: This is an open-label study.

* Preparative Regimen: Patients receive fludarabine IV over 30 minutes on days -7 to -3 and busulfan IV over 2 hours every 6 hours (for a total of 8 doses) on days -4 and -3.
* Graft vs Host Disease (GVHD) Prophylaxis: Patients who have an HLA-identical donor receive oral (or IV if unable to tolerate oral administration) tacrolimus twice daily on days -1 to 90 followed by a taper^* until day 150 and methotrexate IV on days 1, 3, and 6. Patients with a matched related or matched unrelated donor receive oral (or IV if unable to tolerate oral administration) tacrolimus twice daily on days -1 to 180 followed by a taper^* as tolerated; methotrexate IV on days 1, 3, 6, and 11; oral mycophenolate mofetil twice daily on days -2 to 60 followed by a taper; and rabbit anti-thymocyte globulin IV over 4-6 hours on days -4 to -1 (for a total of 4 doses).

NOTE: *Tacrolimus may be tapered on days 60-90 if donor chimerism of CD3+ cells is less than 50% at day 60 or patient has progressive disease

* Allogeneic Stem Cell Transplantation: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on days 0 and 1. Patients then receive filgrastim (G-CSF) subcutaneously daily beginning on day 7 and continuing until blood counts recover.
* Donor Lymphocyte Infusion (DLI): After day 180 (or day 210 for patients without an HLA-identical donor), patients with stable or progressive disease and no active GVHD may receive up to 3 DLIs every 8 weeks.

Patients are followed within 2-3 months, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hematologic malignancy, including one of the following:

  * Chronic lymphocytic leukemia (CLL)

    * Absolute lymphocytosis greater than 5,000/mm^3
    * Lymphocytes must appear morphologically mature with less than 55% prolymphocytes
    * Lymphocyte phenotype with expression of CD19 and CD5
  * Prolymphocytic leukemia (PLL)

    * Morphologically confirmed
    * Absolute lymphocytosis greater than 5,000/mm^3
    * More than 55% prolymphocytes
  * Non-Hodgkin's lymphoma or Hodgkin's lymphoma

    * Any WHO histologic subtype allowed except mantle cell lymphoma
    * Core biopsies allowed if they contain adequate tissue for primary diagnosis and immunophenotyping
    * No bone marrow biopsy as the sole diagnostic means for follicular lymphoma
  * Multiple myeloma

    * Active disease requiring treatment
    * Durie-Salmon stage I, II, or III
  * Acute myeloid leukemia

    * Documented control (i.e., less than 10% bone marrow blasts and no circulating blasts)
  * Myelodysplastic syndromes

    * Documented disease by WHO criteria
* Must have evidence of relapse/progression at least 6 months after prior high-dose chemotherapy with autologous hematopoietic stem cell support
* Absence of CD23 expression for CLL or PLL allowed provided there is no morphologic evidence of mantle cell lymphoma
* Availability of any of the following donor types:

  * HLA-identical sibling (6/6)
  * 9/10 matched related donor by high-resolution molecular typing at HLA A, B, C, DRB1, and DQB1 loci

    * Only a single mismatch at one class I or II allele allowed
  * 10/10 matched unrelated donor by high-resolution molecular typing at HLA A, B, C, DRB1, and DQB1 loci
* No syngeneic donors

PATIENT CHARACTERISTICS:

Age

* Under 70

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal

* Creatinine clearance at least 40 mL/min

Cardiovascular

* LVEF at least 30% by MUGA

Pulmonary

* DLCO greater than 40%
* No symptomatic pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled diabetes mellitus
* No active serious infection
* No known hypersensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior surgery

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2002-12; Primary Completion 2006-11 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality | 6 months post transplant

SECONDARY OUTCOMES:
Per cent donor chimerism | 30, 60, 90, 180 days post transplant
Disease-free survival | 12 months up to 5 years post study entry
Graft-versus-host disease incidence | 6 months post transplant
Response Rates | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Asad Bashey, MD, PhD, Study Chair — University of California, San Diego
Locations (12):
- United States (12):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Bashey A, Owzar K, Johnson JL, Edwards PS, Kelly M, Baxter-Lowe LA, Devine S, Farag S, Hurd D, Ball E, McCarthy P, Lister J, Shea TC, Linker C. Reduced-intensity conditioning allogeneic hematopoietic cell transplantation for patients with hematologic malignancies who relapse following autologous transplantation: a multi-institutional prospective study from the Cancer and Leukemia Group B (CALGB trial 100002). Biol Blood Marrow Transplant. 2011 Apr;17(4):558-65. doi: 10.1016/j.bbmt.2010.07.015. Epub 2010 Jul 30. PMID 20674758
- [Result] Bashey A, Owzar K, Johnson JL, et al.: Reduced-intensity allogeneic transplantation after failure of autologous transplantation: a prospective multi-center CALGB study. [Abstract] Blood 108 (11): A-3122, 2006.